CLINICAL TRIAL: NCT06067750
Title: The Narcotrend Depth of Anaesthesia Monitor as an Indicator of Seizures and Burst Suppression in the Intensive Care Unit
Brief Title: Comparison of Narcotrend and Cerebral Function Analysing Monitor in Intensive Care to Monitor Seizures and Deep Sedation
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 21IT001
Record Dates: First submitted 2023-09-07; First posted 2023-10-05 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage; Intracerebral Haemorrhage; Encephalitis; Acute Ischemic Stroke; Status Epilepticus; Seizures; Subdural Hematoma; ICP (Intracranial Pressure) Increase
Keywords: Narcotrend; Continuous Electroencephalography; Cerebral Function Analysing Monitor; Depth of Anaesthesia Monitor; Seizures; Burst Suppression; Intensive Care
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Cerebral Hemorrhage; Encephalitis; Ischemic Stroke; Status Epilepticus; Seizures; Hematoma, Subdural; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients referred to Clinical Neurophysiology for Cerebral Function Analysing Monitoring (CFAM): Patients referred from both adult and paediatric intensive care units
  Interventions: Diagnostic Test: Narcotrend compared to Cerebral Function Analysing Monitor (CFAM)

INTERVENTIONS:
Diagnostic Test: Narcotrend compared to Cerebral Function Analysing Monitor (CFAM) — All patients will receive Narcotrend and CFAM monitoring in this observational study

SUMMARY:
A study in the use of the Narcotrend depth of anaesthesia monitor to record a) seizures, and b) monitor a level of sedation referred to as 'burst suppression', in sedated patients in the adult and paediatric intensive care.

Studies have shown that patients in coma on the intensive care unit may have subclinical in addition to clinical seizures. Subclinical seizures are seizures that do not show any outward signs and may go undetected.

The current gold standard of recording seizures in the intensive care unit is by non-invasive, continuous monitoring of the electrical activity of the brain by electroencephalography (cEEG) using cerebral function analysing monitor (CFAM).

This is recorded with simultaneous video recording and is performed by Clinical Neurophysiology departments.

There has been a steady increase in demand for this service over recent years. Additionally, CFAM / cEEG is labour intensive and expensive. If trends continue, the proportion of hospitals offering CFAM / cEEG will continue to rise, creating increased demand for specialist staff, of which there are a finite number.

Depth of anaesthesia monitors are used by anaesthetists to assess the level of anaesthesia in sedated patients using specialised, automated EEG analysis and are now recommended by NICE (DG6) to tailor anaesthetic dose to individual patients.

This study aims to investigate the utility of the Narcotrend depth of anaesthesia monitor to monitor for seizures and burst suppression on the adult and paediatric intensive care unit. These monitors are cheaper and more widely available with the scope to be used at every bed space requiring neuro observation on the intensive care unit.

The study aims to recruit all patients who are referred for CFAM / cEEG monitoring at Nottingham University Hospitals (NUH) Trust over a 12 month period. These patients will undergo simultaneous recording using CFAM / cEEG and depth of anaesthesia monitoring.

DETAILED DESCRIPTION:
A non-invasive, prospective, observational, qualitative, comparative study performed on the adult and paediatric intensive care unit of NUH Trust. Study population will be all adult and paediatric patients referred for CFAM monitoring, including, but not limited to patients who are at risk of seizures due to status epilepticus, haemorrhage and traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

Intensive care CFAM is recommended but not confined to identify non-convulsive seizures and non-convulsive status epilepticus (NCSE) in critically ill patients with the following:

1. Persistently abnormal mental status following generalised convulsive status epilepticus (GCSE) or other clinically evident seizures.
2. Acute supratentorial brain injury with altered mental status. This includes traumatic brain injury, subarachnoid hemorrhage, intracerebral hemorrhage, encephalitis, acute ischemic stroke, and during and after therapeutic hypothermia following cardiac arrest.
3. Fluctuating mental status or unexplained alteration of mental status without known acute brain injury: Mental status abnormalities can include agitation, lethargy, fixed or fluctuating neurologic deficits such as aphasia or neglect, obtundation, and coma.
4. Patients requiring pharmacological paralysis and risk for seizures.
5. Clinical paroxysmal events suspected to be seizures, to determine whether they are ictal or non-ictal
6. Patients with suggested secondary brain injury e.g. those with increased intracranial pressure.
7. Monitoring of the response of seizures and status epilepticus to treatment and to a level of burst suppression

Exclusion Criteria:

1. Patients where CFAM has been requested but a routine EEG is thought to be more appropriate, eg. in cases where a routine 20 minute EEG would answer the clinical / referral question.
2. Next of kin will not be approached to consent for the patient to be enrolled into the study where clinical condition dictates that it would not be appropriate eg. imminent withdrawal of care.
3. Participants will be excluded from the study where consent is not granted or withdrawn. This may be at commencement of the study by parents of paediatric patients or next of kin of adult patients.
4. Data gained from patients who regain capacity to give retrospective consent and then withdraw will also be excluded.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be all adult and paediatric patients referred for CFAM monitoring, including, but not limited to patients who are at risk of seizures due to status epilepticus, haemorrhage and traumatic brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Seizure detection | Up to 72 hours monitoring of each patient
  The number of seizures detected and verified by the Narcotrend monitor when compared to the number of seizures detected by conventional CFAM / cEEG monitoring.
  Seizure activity is detected by analysing changes in brain activity. This is done by visually analysing waveforms
Burst suppression monitoring | Up to 72 hours monitoring of each patient
  The number of periods of burst suppression detected and verified by the Narcotrend monitor when compared and detected by conventional CFAM / cEEG monitoring.
  Burst suppression is detected by analysing changes in brain activity. This is done by visually analysing waveforms

SECONDARY OUTCOMES:
Interrater reliability | Up to 72 hours monitoring of each patient
  Compare the interrater reliability between clinical neurophysiology staff and the non-expert reviewers (intensivists / advanced critical care practitioners) in assessing seizures and periods of burst suppression activity using CFAM and Narcotrend equipment.
  The non-expert group will categorise the Narcotrend and CFAM recordings blindly and retrospectively. Their findings will then be compared to clinical neurophysiology findings for the same machines and categories to compare interrater agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Sneath, DClinSci-stu, Principal Investigator — NUH; Ziad Alrifai, MBChB(Hons), Study Director — Nottingham University Hospitals Trust
Locations (1):
- Nottingham University Hospitals Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bader MK, Arbour R, Palmer S. Refractory increased intracranial pressure in severe traumatic brain injury: barbiturate coma and bispectral index monitoring. AACN Clin Issues. 2005 Oct-Dec;16(4):526-41. doi: 10.1097/00044067-200510000-00009. PMID 16269897
- [Background] Arbour RB, Dissin J. Predictive value of the bispectral index for burst suppression on diagnostic electroencephalogram during drug-induced coma. J Neurosci Nurs. 2015 Apr;47(2):113-22. doi: 10.1097/JNN.0000000000000124. PMID 25629593
- [Background] Berger-Estilita J, Steck K, Vetter C, Seidel K, Krejci V, Hight D, Kaiser H. A case report of several intraoperative convulsions while using the Narcotrend monitor: Significance and predictive use. Medicine (Baltimore). 2019 Nov;98(47):e18004. doi: 10.1097/MD.0000000000018004. PMID 31764814
- [Background] Dahaba AA, Liu DW, Metzler H. Bispectral index (BIS) monitoring of acute encephalitis with refractory, repetitive partial seizures (AERRPS). Minerva Anestesiol. 2010 Apr;76(4):298-301. PMID 20332745
- [Background] Dwivedi D, Bhatnagar V, Kiran S, Ray A. Intraoperative seizures during redo cranioplasty for sinking skin flap syndrome- Role of BIS monitor in detection. Saudi J Anaesth. 2017 Jul-Sep;11(3):359-360. doi: 10.4103/sja.SJA_44_17. No abstract available. PMID 28757846
- [Background] Iturri Clavero F, Tamayo Medel G, de Orte Sancho K, Gonzalez Uriarte A, Iglesias Martinez A, Martinez Ruiz A. Use of BIS VISTA bilateral monitor for diagnosis of intraoperative seizures, a case report. Rev Esp Anestesiol Reanim. 2015 Dec;62(10):590-5. doi: 10.1016/j.redar.2015.03.006. Epub 2015 May 3. PMID 25944463
- [Background] Tallach RE, Ball DR, Jefferson P. Monitoring seizures with the Bispectral index. Anaesthesia. 2004 Oct;59(10):1033-4. doi: 10.1111/j.1365-2044.2004.03953.x. No abstract available. PMID 15488073